CLINICAL TRIAL: NCT00503789
Title: The Effect of Infant Feeding on Stool Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Deolinda Scalabrin, Mead Johnson
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 33715
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
Keywords: Healthy infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): cow-milk based infant formula
  Interventions: Procedure: fecal bacteria analysis
- 2 (Experimental): cow milk based infant formula with prebiotics
  Interventions: Procedure: fecal bacteria analysis
- 3 (Other): human milk reference group
  Interventions: Procedure: fecal bacteria analysis

INTERVENTIONS:
Procedure: fecal bacteria analysis — ad lib feeding

SUMMARY:
Infants will be fed infant formula and stool characteristics assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term infants
* 21-30 days of age

Exclusion Criteria:

* Infants with feeding difficulties
* Use of antibiotics or steroids

Ages: 21 Days to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
fecal bacteria analysis | 60 days

SECONDARY OUTCOMES:
Intake, tolerance, stool characteristics, anthropometrics | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Deolinda Scalabrin, MD, Study Director — Mead Johnson Nutrition
Locations (23):
- United States (23):
  - Central Arkansas Pediatric Clinic, Benton, Arkansas
  - Arkansas Pediatrics of Conway, Conway, Arkansas
  - The Children's Clinic of Jonesboro, Jonesboro, Arkansas
  - Altamonte Pediatric Associates, Altamonte Springs, Florida
  - Advocate Center for Pediatric Research, Park Ridge, Illinois
  - Internal Medicine and Pediatrics, Fishers, Indiana
  - East Washington Pediatrics, Indianapolis, Indiana
  - Children's Hospital of Iowa, Coralville, Iowa
  - University of Kansas Medical University, Kansas City, Kansas
  - PTCU/Children and Youth Project, Louisville, Kentucky
  - ACC Pediatric Research, Bossier City, Louisiana
  - ProMed Healthcare, Kalamazoo, Michigan
  - ProMed Pediatrics, Portage, Michigan
  - ProMed Physicians-Pediatrics, Richland, Michigan
  - The Center for Human Nutrition, Omaha, Nebraska
  - Winthrop Pediatric Associates, Mineola, New York
  - Cary Pediatric Center, P.A., Cary, North Carolina
  - Pediatric Associates of Mt. Carmel, Inc., Cincinnati, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Northeast Cincinnati Pediatric Assoc, Mason, Ohio
  - Red Lion Pediatrics, Philadelphia, Pennsylvania
  - Alpha Clinical Research, Clarksville, Tennessee
  - Austin Diagnostic Clinic, Austin, Texas

REFERENCES:
- [Derived] Salminen S, Endo A, Isolauri E, Scalabrin D. Early Gut Colonization With Lactobacilli and Staphylococcus in Infants: The Hygiene Hypothesis Extended. J Pediatr Gastroenterol Nutr. 2016 Jan;62(1):80-6. doi: 10.1097/MPG.0000000000000925. PMID 26230902
- [Derived] Scalabrin DM, Mitmesser SH, Welling GW, Harris CL, Marunycz JD, Walker DC, Bos NA, Tolkko S, Salminen S, Vanderhoof JA. New prebiotic blend of polydextrose and galacto-oligosaccharides has a bifidogenic effect in young infants. J Pediatr Gastroenterol Nutr. 2012 Mar;54(3):343-52. doi: 10.1097/MPG.0b013e318237ed95. PMID 21946836